CLINICAL TRIAL: NCT02431949
Title: A Cross-sectional Analysis of Musical Ability in Patients With Refractory Schizophrenia
Brief Title: The Music Study in Refractory Psychosis
Acronym: MARS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H14-02891
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Schizophrenia; Psychosis
Keywords: Music; Amusia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: Participants without a psychosis disorder diagnosis.
- Patients: Participants with a psychosis disorder diagnosis- recruited from the BC Psychosis Program.
  Interventions: Other: Admission to BCPP

INTERVENTIONS:
Other: Admission to BCPP — There is no intervention associated with this study.
  Groups: Patients

SUMMARY:
The perception of music requires coordinated neural activities in distributed multi-functional centers across both hemispheres. The association between musical abilities and other general cognitive functions have been studied in several populations with inconsistent results.

Schizophrenia is a major mental disorder that is strongly associated with cognitive deficits. These often appear before the onset of psychotic symptoms and persist throughout effective treatment of positive and negative symptoms. Like other disorders of psychosis, schizophrenia features general deficits in auditory memory and sensory processing. Recently, Sawada et al. (2014) and Wen et al. (2014) studied music abilities in Japanese and Chinese schizophrenic populations. They both used a standardized assessment for amusia called Montreal Battery of Evaluation of Amusia (MBEA) and found marked impairments in perception of scale, contour, interval, rhythm, meter and memory. Both studies showed that deficits in music perception were associated with cognitive deficits and negative symptoms. In regards to positive symptoms, Wen et al., but not Sawada et al., found a significant association.

The present clinical study will assess musical abilities using the MBEA in a Canadian population with and without refractory psychosis. It will explore associations between musical deficits, positive and negative psychiatric symptomology and cognition. The patient population will have a diagnosis of schizophrenia, schizoaffective disorder, affective disorder with psychosis or non substance-related psychosis who were referred to the British Columbia Psychosis Program (BCPP) due to inadequate or no response to at least two trials of antipsychotics. A focus on refractory psychosis may provide greater insights because these patients have relatively more pronounced psychiatric symptoms and cognitive deficits. It will also be valuable to administer the MBEA assessment on a Canadian population, because the test was originally intended for Western populations and its musical phrases were designed with Western tonalities.

DETAILED DESCRIPTION:
1. BACKGROUND, PURPOSE AND JUSTIFICATION

   The perception of music requires coordinated neural activities in distributed multi-functional centers across both hemispheres. The association between musical abilities and other general cognitive functions have been studied in several populations with inconsistent results.

   Schizophrenia is a major mental disorder that is strongly associated with cognitive deficits. These often appear before the onset of psychotic symptoms and persist throughout effective treatment of positive and negative symptoms. Like other disorders of psychosis, schizophrenia features general deficits in auditory memory and sensory processing. Recently, Sawada et al. (2014) and Wen et al. (2014) studied music abilities in Japanese and Chinese schizophrenic populations. They both used a standardized assessment for amusia called Montreal Battery of Evaluation of Amusia (MBEA) and found marked impairments in perception of scale, contour, interval, rhythm, meter and memory. Both studies showed that deficits in music perception were associated with cognitive deficits and negative symptoms. In regards to positive symptoms, Wen et al., but not Sawada et al., found a significant association.

   The present clinical study will assess musical abilities using the MBEA in a Canadian population with and without refractory psychosis. It will explore associations between musical deficits, positive and negative psychiatric symptomology and cognition. The patient population will have a diagnosis of schizophrenia, schizoaffective disorder, affective disorder with psychosis or non substance-related psychosis who were referred to the British Columbia Psychosis Program (BCPP) due to inadequate or no response to at least two trials of antipsychotics. A focus on refractory psychosis may provide greater insights because these patients have relatively more pronounced psychiatric symptoms and cognitive deficits. It will also be valuable to administer the MBEA assessment on a Canadian population, because the test was originally intended for Western populations and its musical phrases were designed with Western tonalities.
2. RESEARCH OUTLINE This is a cross-sectional, observational study. Participating patients with refractory psychosis and healthy (age- and gender- matched) controls will undergo the Montreal Battery of Evaluation of Amusia assessment and assessments of cognition and symptoms.

The purpose of the study is to describe music perceptive ability in patients with refractory psychosis using the Montreal Battery of Evaluation of Amusia, a standardized and continuous measure of musical ability. The criterion for amusia is a score of 2 standard deviations below the mean of normal participants.

4) OBJECTIVES

Primary:

The primary objective is to compare music perceptive ability in patients with clinically identified refractory psychosis with healthy subjects.

Secondary:

The secondary objectives are to compare the prevalence of amusia in a population of patients with refractory psychosis versus a population of healthy controls, and to compare psychiatric symptoms and cognition in patients with amusia versus patients without amusia. We will also determine if an association exists between music perceptive ability and:

* General and specific aspects of symptom severity, as assessed by standardized symptom rating scales and neurological status examination.
* General and specific aspects of cognition, as assessed by cognitive tests.
* Demographic variables such as sex, age, musical training and education. In addition, we will investigate potential pathways between symptomologies of psychosis, cognitive deficits and musical disability (if found) by using exploratory mediation analysis.

  5) RESEARCH METHOD We will recruit 100 participants, who will undergo the Montreal Battery of Evaluation of Amusia test and cognitive tests. Of these, 50 will be age- and gender- matched participants not diagnosed with a psychosis disorder who will serve as controls. The remaining 50 participants will be recruited from BCPP at UBC Hospital for in-patients diagnosed with refractory psychosis. For patients, participation will also involve assessments of their mental health (psychiatric symptoms).

  6) STATISTICAL ANALYSIS Inferential analyses will be used to assess differences in musical ability between patients and controls. It will also be used to evaluate differences in psychiatric symptoms and cognition between patients with amusia and those without amusia. Linear regression analyses will be done to relate psychiatric symptoms and cognition to musical ability. Mediation analyses will be performed to determine a causal model between symptoms, cognition and musical ability.

ELIGIBILITY:
Inclusion Criteria:

* Admission to BC Psychosis Program at UBC Hospital in Vancouver, B.C. with a diagnosis of a psychosis disorder (patients only)
* Fluency in English (patients and controls)
* Able to give consent

Exclusion Criteria:

For controls and patients:

• Presence of hearing deficits

For controls only, history of:

* Diagnosis of psychosis disorder
* Antipsychotic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participant population will include all patients who have been admitted to the British Columbia Psychosis Progarm (BCPP) at the University of British Columbia (UBC) Hospital. Admission criteria to BCPP include the following: 1) Must be 18 years or older who are medically stable; 2) Diagnosis of schizophrenia, schizoaffective disorder, mood disorder with psychosis, or non-substance-related psychosis requiring diagnostic clarification; 3) History of no response or inadequate response of positive symptoms to at least 2 adequate trials of antipsychotics (one of which is a second generation agent) by health authority tertiary clinical teams; 4) Incomplete recovery of social, vocational, and occupational functioning likely to respond to active intervention. Control subjects will be age and gender matched with patient participants.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Musical Ability (The Montreal Battery of Evaluation of Amusia) | 2 hours
  Assessment of musical ability based on scores from The Montreal Battery of Evaluation of Amusia

SECONDARY OUTCOMES:
Cognitive Ability (NIH toolbox-cognitive battery scores) | 1 hour
  NIH toolbox-cognitive battery scores.
Mental Health Symptom Severity (Rating scales from Sci-PANSS and MINI Neuropsychiatric Interview) | 2 hours
  Rating scales from Sci-PANSS and MINI Neuropsychiatric Interview.

CONTACTS AND LOCATIONS:
Overall Officials: Alasdair Barr, PhD, Principal Investigator — The University of British Columbia
Locations (1):
- BC psychosis ward at UBC Hospital, Vancouver, British Columbia, Canada